CLINICAL TRIAL: NCT05396716
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Postoperative Nausea and Vomiting After Liver Surgery
Brief Title: Acupoint Stimulation Alleviates Postoperative Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XJH-A-20220410
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: PONV
Keywords: transcutaneous electrical acupoint stimulation; liver surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The stimulator is put in an opaque box
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical acupoint stimulation (Experimental)
  Interventions: Device: transcutaneous electrical acupoint stimulation
- Control (No Intervention)

INTERVENTIONS:
Device: transcutaneous electrical acupoint stimulation — Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given during surgery.
  Other Names: TEAS
  Arms: transcutaneous electrical acupoint stimulation

SUMMARY:
Incidence of postoperative nausea and vomiting (PONV) could be high as 60% after liver surgery. Acupoint stimulation has been proved to decrease PONV. In this study, we will investigate the effect of transcutaneous electrical acupoint stimulation on incidence of PONV after liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* scheduled for elective liver surgery under general anesthesia

Exclusion Criteria:

* body mass index less than 18 kg/m2 or higher than 30 kg/m2
* American Society of Anesthesiologists status higher than Ⅲ
* patients with contraindication to transcutaneous electrical stimulation, including skin damage, infection or implantable electrical device
* suspected or existed abuse of drug or alcohol
* pregnant or breeding women
* history of neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
incidence of nausea and vomiting by 24 hours after surgery | from end of surgery to 24 hours after surgery, in a total of 24 hours

SECONDARY OUTCOMES:
incidence of nausea and vomiting by 48 hours after surgery | from end of surgery to 48 hours after surgery, in a total of 48 hours
incidence of nausea and vomiting in PACU (post-anesthesia care unit) | from end of surgery to discharge from PACU(post-anesthesia care unit), in an average of 30 minutes
score of nausea and vomiting by 24 hours after surgery | from end of surgery to 24 hours after surgery, in a total of 24 hours
score of nausea and vomiting by 48 hours after surgery | from end of surgery to 48 hours after surgery, in a total of 48 hours
score of nausea and vomiting in PACU(post-anesthesia care unit) | from end of surgery to discharge from PACU, in an average of 30 minutes
Quality of recovery score at 24 hours after surgery | from end of surgery to 24 hours after surgery, in a total of 24 hours
Quality of recovery score at 48 hours after surgery | from end of surgery to 48 hours after surgery, in a total of 48 hours
postoperative in-hospital stay | from end of surgery to discharge from hospital, in an average of 7 days
death by 6 months after surgery | from end of surgery to 6 months after surgery, in a total of 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee A, Chan SK, Fan LT. Stimulation of the wrist acupuncture point PC6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2015 Nov 2;2015(11):CD003281. doi: 10.1002/14651858.CD003281.pub4. PMID 26522652